CLINICAL TRIAL: NCT00521573
Title: Effects of Chocolate on Coronary Vasomotion in Patients After Heart Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: EK1129
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dark chocolate

SUMMARY:
The aim of the present study is to investigate whether the ingestion of a flavonoid-rich dark chocolate compared to flavonoid-free placebo chocolate will improve coronary vasomotion in heart transplanted patients.

DETAILED DESCRIPTION:
Dark chocolate contains a high amount of flavonoids. Flavonoids hold the possibilities to improve oxidative stress and hence the possibility to improve endothelium-dependent coronary vasomotion, which is a powerful surrogate for clinical prognosis. Coronary atherosclerosis is promoted by impaired endothelial function and increased platelet activation. High oxidative stress and reduced antioxidant defenses play a crucial role in the pathogenesis of atherosclerosis, in particular in transplanted hearts. The aim of the present study is to investigate whether the ingestion of a flavonoid-rich dark chocolate compared to flavonoid-free placebo chocolate will improve coronary vasomotion in heart transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients after heart transplantation not requiring immediate coronary intervention
2. Age 20 - 80
3. Written obtained informed consent

Exclusion Criteria:

1. Heart failure (acute or chronic >NYHA II)
2. Ventricular tachy-arrythmias or AV-Block >I°
3. Renal insufficiency (>200 μmol/l) or liver disease (ALT or AST >150 IU)
4. Symptomatic hypotension, hypertension >160/100mmHg
5. Known allergy to compounds dark chocolate
6. Acute infectious disease
7. Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
8. Participation in another study within the last month
9. Concomitant vitamin supplements

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corti, MD, Principal Investigator — University of Zurich